CLINICAL TRIAL: NCT02828891
Title: Analysis of Translaminar Pressure Gradient Using Noninvasive Cerebrospinal Fluid Pressure Monitoring
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: This study is being closed due to the inability to acquire the required technology to complete the study
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Richard K. Lee, Associate Professor of Ophthalmology, Cell Biology and Neuroscience, University of Miami
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 20160505
Record Dates: First submitted 2016-07-01; First posted 2016-07-12 (Estimated); Last update posted 2020-10-30 (Actual); Status verified 2020-10

CONDITIONS: Glaucoma
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Experimental (Experimental): Intervention: transcranial Doppler device will be utilized to measure CSF pressure.
  Interventions: Device: Two-Dimensional Transcranial Doppler

INTERVENTIONS:
Device: Two-Dimensional Transcranial Doppler — Transcranial Doppler will be used to measure CSF pressure.

SUMMARY:
This is a single center, prospective study to calculate cerebrospinal fluid pressure (CSFp) using a non-invasive device and assess its role in the development of optic neuropathy due to glaucoma or idiopathic intracranial hypertension (IIH). The study also aims to assess whether CSFp differs between untreated and treated patients with glaucoma, ocular hypertension, IIH, and other ocular diseases that may be associated with CSFp differences.

DETAILED DESCRIPTION:
The pathophysiology of primary open-angle glaucoma (POAG) remains unclear, with potentially a multifactorial etiology. Intraocular pressure (IOP) is the only known modifiable risk factor, yet two clinical conundrums remain - patients with elevated IOP who do not develop glaucoma (ocular hypertension, OHTN) as well as patients with IOP <21 mmHg who still develop glaucoma (normal tension glaucoma, NTG). The etiology of these two scenarios remains unclear.

The role of cerebrospinal fluid pressure (CSFp) in glaucomatous optic neuropathy was initially raised 30-40 years ago. This concept has garnered more interest recently due to new findings in this area. Patients who underwent lumbar puncture (LP) and had POAG were found to have lower CSFp compared to controls in a chart review. Further studies demonstrated a positive correlation between optic nerve damage and the translaminar pressure gradient (TPG), calculated as the CSFp subtracted from the IOP. In 2010, a Chinese group suggested that normal-tension glaucoma (NTG) patients have significantly lower CSFp compared to POAG, and that TPG is greater in NTG and POAG patients compared to controls. The same group also showed that OHTN patients have higher CSFp than POAG patients, suggesting a protective effect of high CSFp when IOP is elevated. Thus, a role for CSFp in the pathophysiology of glaucoma may exist.

One can consider IIH as a model for these forms of glaucoma; CSFp is elevated in IIH, as measured by lumbar puncture (LP). Visual field loss in this disease follows an arcuate pattern, similar to glaucomatous loss. This would seem to suggest that glaucomatous optic neuropathy and IIH optic neuropathy share similar mechanisms (i.e., increased TPG due to either elevated IOP or CSFp).

One of the main hindrances to testing these hypotheses further has been the invasive nature of LP, which involves inserting a large-bore needle into the spinal column. This procedure has a relatively high risk of complications given its proximity to the spinal cord and the potential for traumatic nervous system injury if improperly performed. In contrast to this invasive procedure, a non-invasive computational device was recently developed and CE mark approved to measure CSFp using a two-depth transcranial Doppler device (TDTCD). The underlying principle of the device involves the ophthalmic artery. When originating from the internal carotid artery, the ophthalmic artery is within the subarachnoid space and thus is mildly compressed by CSFp. After exiting the intracranial space into the orbit, the ophthalmic artery loses its subarachnoid surrounding, and is no longer affected by CSFp. The TDTCD applies minimal external pressure to the orbit such that the pressure exerted externally on the extracranial segment is equivalent to the CSFp exerted on the intracranial segment (as measured by Doppler signals of both vessels.) The safety of the device has been demonstrated and verified; it has obtained CE certification in Europe, and is currently awaiting FDA approval with a "Non-Significant Risk" categorization. Further details regarding the device can be viewed at www.vittamed.com.

The device has been shown to correlate extremely well with the gold standard of LP. Multiple clinical trials utilizing this device in noninvasive CSFp monitoring in neurosurgical patients are underway at various other institutions, including Johns Hopkins University, NASA, and Baylor College of Medicine.

The investigators propose utilizing TDTCD to non-invasively measure CSFp in glaucoma/OHTN patients, IIH patients, and controls at various stages in treatment in order to further delineate the possible role of TPG in the pathophysiology of these conditions. The investigators believe this non-invasive approach has the potential to alter our current understanding and management of these disease processes, thereby assisting in the identification of at-risk patients more accurately, improving patients' quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Open angle with normal structures on gonioscopy
* Patients with a diagnosis of, or at risk for the development of, optic neuropathy, including NTG, POAG, OHTN, IIH (in addition to controls)

Exclusion Criteria:

* Known abnormal vascular anatomy (i.e., abnormal anatomy of the ophthalmic artery)
* Alzheimer's disease or other neurodegenerative diseases
* Known abnormal intracranial anatomy or malformations
* Minors, prisoners, pregnant patients
* Patients unable to consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-07; Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Mean CSFp for all groups and controls at various time points (e.g., prior to and after medical or surgical intervention) in order to assess for significant differences. | The investigators anticipate to enroll the subjects over a period of 12 months. The estimated time required for data analysis is 6 months following enrollment of all subjects.
  CSF pressure

SECONDARY OUTCOMES:
Translaminar pressure gradient (calculated as IOP - CSFp) for all groups and controls at various time points (e.g., prior to and after medical or surgical intervention) in order to assess for significant differences. | The investigators anticipate to enroll the subjects over a period of 12 months. The estimated time required for data analysis is 6 months following enrollment of all subjects.
  CSF pressure

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Berdahl JP, Fautsch MP, Stinnett SS, Allingham RR. Intracranial pressure in primary open angle glaucoma, normal tension glaucoma, and ocular hypertension: a case-control study. Invest Ophthalmol Vis Sci. 2008 Dec;49(12):5412-8. doi: 10.1167/iovs.08-2228. Epub 2008 Aug 21. PMID 18719086
- [Background] Berdahl JP, Allingham RR, Johnson DH. Cerebrospinal fluid pressure is decreased in primary open-angle glaucoma. Ophthalmology. 2008 May;115(5):763-8. doi: 10.1016/j.ophtha.2008.01.013. PMID 18452762
- [Background] Ren R, Jonas JB, Tian G, Zhen Y, Ma K, Li S, Wang H, Li B, Zhang X, Wang N. Cerebrospinal fluid pressure in glaucoma: a prospective study. Ophthalmology. 2010 Feb;117(2):259-66. doi: 10.1016/j.ophtha.2009.06.058. Epub 2009 Dec 6. PMID 19969367
- [Background] Ren R, Zhang X, Wang N, Li B, Tian G, Jonas JB. Cerebrospinal fluid pressure in ocular hypertension. Acta Ophthalmol. 2011 Mar;89(2):e142-8. doi: 10.1111/j.1755-3768.2010.02015.x. PMID 21348961
- [Background] Ragauskas A, Matijosaitis V, Zakelis R, Petrikonis K, Rastenyte D, Piper I, Daubaris G. Clinical assessment of noninvasive intracranial pressure absolute value measurement method. Neurology. 2012 May 22;78(21):1684-91. doi: 10.1212/WNL.0b013e3182574f50. Epub 2012 May 9. PMID 22573638